CLINICAL TRIAL: NCT02259712
Title: Effectiveness of Hypopressive Exercises Versus Pelvic- Perineal Physiotherapy in Women With Pelvic Floor Dysfunction: Randomised, Single-blinded, Clinical Trial.
Brief Title: Effectiveness of Hypopressive Exercises Versus Pelvic-perineal Physiotherapy
Acronym: HEPFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Beatriz Navarro Brazález, Physical Therapy researcher, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OE 20/2013; OE 20/2013 (Other: Ethics Committee of University Hospital Prince of Asturias)
Record Dates: First submitted 2014-09-05; First posted 2014-10-08 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Pelvic Floor Disorders; Urinary Incontinence; Fecal Incontinence; Pelvic Pain
Keywords: Women; Pelvic floor disorders; Urinary incontinence; Fecal incontinence; Physical Therapy Modalities
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence; Fecal Incontinence; Pelvic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pelvic-perineal physiotherapy (Active Comparator): The treatment duration is 2 days per week during 8 weks (two months). The aproximate duration of the season is 45 minutes. The protocol consists in:
  1. Anatomical and physiological explanation of the pelvic girdle (perineal organs bony, ligaments and muscular structures of the entire abdominal and pelvic cavity).
  2. Hygienic and behavioral advises preventing pelvic floor dysfunctions.
  3. Awareness of the pelvic floor muscles.
  4. Strengthening the pelvic floor muscles and the entire abdominal pelvic cavity. Use of electrostimulation and biofeedback in different positions if deemed necessary.
  5. Treatment the abdominal-pelvic cavity pain if it requires.
  Interventions: Behavioral: Therapeutic education.; Other: Pelvic-perineal physiotherapy; Other: Physical Therapy assessment
- Hyporessive and Pelvic-perineal PT (Experimental): The treatment duration is 2 days per week, 8 weeks (two months). The session is about 45 minutes. All women are instructed on hygienic and behavioral advises preventing pelvic floor dysfunctions. They are teach basic anatomy and physiology to understand the importance of these advises and anatomical and physiological explanation of the pelvic girdle. The participants are also treated by doing Hypopressive exercises and by specific physiotherapy for the strengthening the pelvic floor muscles.
  Interventions: Other: Hypopressive exercises; Behavioral: Therapeutic education.; Other: Pelvic-perineal physiotherapy; Other: Physical Therapy assessment
- Hypopressive exercises (Experimental): The treatment is done 2 times per week for 8 weeks (2 months). The session duration is about 45 minutes. All participants are instructed on hygienic and behavioral advises preventing pelvic floor dysfunctions. They are teach basic anatomy and physiology to understand the importance of these advises and anatomical and physiological explanation of the pelvic girdle (perineal organs bony, ligaments and muscular structures of the entire abdominal and pelvic cavity). The participants are also treated by doing Hypopressive exercises in standing, sitting, and supine fours.
  Interventions: Other: Hypopressive exercises; Behavioral: Therapeutic education.; Other: Physical Therapy assessment

INTERVENTIONS:
Other: Hypopressive exercises — 45 minutes treatment by hipopressive exercises 2 times per week during 8 weeks. They will be doing in different positions: standing, kneeling, sitting and lying. The patient will be teach a total of 30 exercises. In the week number 8 the women with the physical therapist will choose 3 exercises that will be done daily at home during 20 minutes.
  Other Names: Hypopressive kinesiotherapy
  Arms: Hypopressive exercises; Hyporessive and Pelvic-perineal PT
Behavioral: Therapeutic education. — The therapeutic education will be doing during the 8 weeks of treatment. In the first day the knowledge and the briefs of the pelvic floor dysfunction will be assessed. Dietary and behavioral habits will also be discussed. In the second day anatomical and physiological explanation of the pelvic girdle will be the priority. In the third day will be explained the signs and symptoms of the different pelvic floor dysfunctions. In the four day will be analyzed the risk factors that may cause or worsen pelvic floor dysfunctions.
  In the fifth day will be begun to correct the bad habits. In the last day will be reviewed the knowledge and new habits acquired during the treatment. In all treatment days will be discussed the doubts of the participant.
  Other Names: Hygienic and behavioral advises.
Other: Pelvic-perineal physiotherapy — 45 minutes physical therapy treatment 2 times per week during 8 weeks. There will be done specific exercises of the pelvic floor muscles and coordination exercises of the pelvic floor muscles with other muscles in different positions. Electrostimulation, biofeedbak, cones and dinamometric devices can be employed to improve the muscle performance.
  Other Names: Specific physical therapy.
  Arms: Hyporessive and Pelvic-perineal PT; Pelvic-perineal physiotherapy
Other: Physical Therapy assessment — Pre-treatment, post-treatment, 3, 6 and 12 months after physical therapy treatment. Will be done a specific evaluation of pelvic floor muscles using the Modified Oxford Scale, superficial electromyography, perineometry and dynamometer. For the evaluation of the impact, the signs and the symptoms questionnaires will be completed by the participants.
  Other Names: Physiotherapy evaluation

SUMMARY:
Introduction: Hypopressive Exercises are included within a method of physiotherapy which was created with the purpose of strengthening the deep muscles of the abdomen without damaging ligamentous and muscular structures of the perineum, also strengthening the muscles of pelvic floor reflexively. Although this technique has been included as treatment and a prevention method of pelvic floor dysfunction, there are few studies supporting its benefits. The investigators hypothesis is that the combination of both physiotherapy treatments will provided the best results for women who suffer pelvic floor dysfunctions.

Objective: To determine whether Hypopressive Exercises are an option to include in the physiotherapy treatment of women suffer at least one pelvic floor dysfunction and whether the results reported are comparable to those provided by pelvic-perineal physiotherapy.

Subjects and methods: A randomized clinical trial, the examiner being blinded unaware of the intervention group to which subjects were assigned. Participants will be randomly assigned to three groups:

1. An experimental group, where the participants will be treated by Hypopressive exercises and hygienic and behavioral measures;
2. Another experimental group where pelvic-perineal physiotherapy will join with Hypopressive exercises and hygienic and behavioral advises;
3. And a third group where will be done pelvic-perineal physiotherapy and hygienic and behavioral measures.

Pre- intervention, immediate post-intervention, 3, 6 and 12 months assessments will be made. The selection criteria will be: adult women who present signs and symptoms that indicate a pelvic floor dysfunction or have a medical diagnosis to confirm it. All participants must understand and sign freely Informed Consent.

Sample size: Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 26 subjects were required in each group to detect a difference equal to or greater than 3 microvolts (Total of 78 subjects). It assumes a standard deviation of 4.8 microvolts and the rate of loss to follow up esteem 20% (Magalhães-Resende et al. 2012).

Data Analysis: A descriptive analysis of all variables was performed. It establish for all cases a confidence level of 95% (p <0.05). The effectiveness was assessed by comparing the experienced change of the three goups in outcome variables between physicaltherapy examinations.

ELIGIBILITY:
Inclusion Criteria:

* Women who experience signs and symptoms evidencing pelvic floor dysfunction.
* Women with a medical diagnosis of pelvic floor dysfunction.
* Women with signs and or symptoms of urinary incontinence, anal incontinence, overactive bladder syndrome and prolapse in grade I-II.
* All participants must understand and sign freely Informed Consent.

Exclusion Criteria:

* Women minors.
* Pregnant women.
* Women who have had a vaginal delivery or cesarean in the past six months.
* Women with pelvic floor dysfunction which is serious and the first indication is surgical (prolapses grades III-IV).
* Women who have been treated for perineal physiotherapy in the past 12 months.
* Participants submit any pathology that may affect treatment (neurological, gynecological or urological), or recurrent urinary tract infection or hematuria.
* Women with cognitive limitations in understanding the information, respond to questionnaires, consent and / or participate in the study.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
The change of signs, symptoms and impact of pelvic floor dysfunction between reviews | Pre-treatment, post-treatment, 3, 6 and 12 months assessments were required.
  - Improve the impact of pelvic floor dysfunctions by 30% according to Spanish short version of Pelvic Floor Impact Questionnaire (PFIQ-7).
The change of signs, symptoms and impact of pelvic floor dysfunction between reviews | Pre-treatment, post-treatment, 3, 6 and 12 months assessments were required.
  - Improve the signs and symptoms of pelvic floor dysfunction by 30% according to Spanish short version of Pelvic Floor Distress Inventory (PFDI-20).

SECONDARY OUTCOMES:
The change of pelvic floor muscles strenght | Pre-treatment, post-treatment, 3, 6 and 12 months assessments were required.
  - Improve the strength of the pelvic floor muscles by 2 points according to the Modified Oxford Scale.
The change of pelvic floor muscles pressure force | Pre-treatment, post-treatment, 3, 6 and 12 months assessments were required.
  - Improve the strength of pelvic floor in 10 cm H2O measured with digital perineometer.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz N Navarro, PhD student, Principal Investigator — University of Alcala
Locations (1):
- Teacher care and research in physiotherapy Unit. Department of Physiotherapy. University of Alcala., Alcalá de Henares, Madrid, Spain

REFERENCES:
- See also: Women's Health Research Group Info — https://fisioterapia-saludmujer.web.uah.es/